CLINICAL TRIAL: NCT04753632
Title: Assessment of the Biopsychosocial Status of People With Cerebral Palsy and Related Diseases and Their Caregivers During the COVID-19 Pandemic
Brief Title: Status of People With Cerebral Palsy and Their Caregivers During COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator; PT; PhD, Universidad de Granada
Other Study IDs: DF0095UG
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral palsy patients and caregivers: Cerebral palsy patients and caregivers
- Healthy people and their caregivers: Healthy people and their caregivers

SUMMARY:
COVID-19, as well as the collateral situations that it entails, has been causing panic, anguish and anxiety that has generated biopsychosocial problems in society affecting not only the physical and social level but also the mental health and well-being.

The main objective of this research project is to assess the biopsychosocial status of people with cerebral palsy and related diseases and their caregivers during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy patients and their caregivers

Exclusion Criteria:

* Patients or caregivers with Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cerebral palsy patients and their caregivers
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Questionnaire of Knowledge, attitudes and practice towards COVID-19 | Baseline
  Questionnaire to evaluate the knowledge about COVID-19. It includes 12 items. Patients have to answer true/false. Higher puntuation indicates better knowledge results.
Caregiver COVID-19 limitation scale | Baseline
  This scale is used to examine the impact of the COVID-19 pandemic on caregivers. Scores ranged from 1 to 10, and a higher score indicates more limitations.
Fear of Coronavirus-19 Scale | Baseline
  It is a scale that assesses the fear of COVID-19. It consists of 7 items scored on a 5-item Likert scale. The higher the score, the more fear.
Covid-19 Stress Scale (CSS) | Baseline
  COVID stress scale (CSS): is a 36-item COVID Stress Scale (CSS) to measure these features, as they pertain to COVID-19. The CSS were developed to better understand and assess COVID-19-related distress. The scales were intentionally designed so they could be readily adapted for future pandemics.
Coronavirus Anxiety Scale (CAS) | Baseline
  Coronavirus anxiety scale (CAS): It is a scale that measures the anxiety generated by COVID-19 in the last two weeks.
  It presents 5 items and a score> 9 indicates dysfunctional anxiety associated with the pandemic.
Connor-Davidson Resilience Scale-10 | Baseline
  Connor-Davidson Resilience Scale (CD-RISC) was used to measure resilience. Respondents are asked to answer on a five-point Likert scale (0 = totally disagree to 4 = totally agree)
COPE | Baseline
  The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. "Coping" is defined broadly as an effort used to minimize distress associated with negative life experiences
Medical Outcomes Study-Social Support Survey | Baseline
  This brief, self-administered Social Support Survey instrument was developed for patients in the Medical Outcomes Study (MOS), a two-year study of patients with chronic conditions. Higher puntuations indicate higher social support.
Zarit Burden Inventory | Baseline
  The Zarit Burden Inventory examines burden associated with functional/behavioural impairments and the home care situation. Higher puntuations indicate higher burden.

SECONDARY OUTCOMES:
Euroqol-5D | Baseline
  The perception of the level of health and the quality of life were evaluated with the questionnaire European Quality of
  Life-5 Dimensions (EQ-5D). It is composed of 2 parts in which health status is assessed:
  Descriptive system: It consists on 5 dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients classify their health status in 3 severity levels: having no problems, having some or moderate problems, being unable to do/having extreme problems. Visual Analog Scale, by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status)
Hospital Anxiety and Depression Scale | Baseline
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS) . This scale is composed of 14 items divided into two subscales, 7 items of anxiety and 7 items of depression, involving higher values worse psycho-emotional state.
Pittsburgh Sleep Quality Index | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances in the previous month.
International Physical Activity Questionnaire | Baseline
  The International Physical Activity Questionnaire (IPAQ) was developed to measure health-related physical activity (PA) in populations. Higher scores indicates higher physical activity levels.
Functional independence measure | Baseline
  The Functional Independence Measure (FIM) is an 18-item measurement tool that explores an individual's physical, psychological and social function. Higher scores mean a better outcome.
Gross motor function classification system | Baseline
  The GMFCS, or Gross Motor Function Classification System, is a five-level classification that differentiates children with cerebral palsy based on the child's current gross motor abilities, limitations in gross motor function, and need for assistive technology and wheeled mobility.
Manual Agility Classification System | Baseline
  The Manual Ability Classification System (MACS) describes how children with cerebral palsy use their hands to handle objects in daily activities. MACS describes five levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: No